CLINICAL TRIAL: NCT06466460
Title: Motion-based Interactive Technology for Improved Quality of Life in Individuals With Cognitive Impairment
Acronym: WakeIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marie Matérne (Other)
Collaborators: Region Örebro County (Other)
Responsible Party: Sponsor-Investigator, Marie Matérne, Associate professor, Örebro University, Sweden
Organization: Örebro University, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wake it _OrebroU
Record Dates: First submitted 2024-06-07; First posted 2024-06-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Cognitive Impairment
Keywords: interactive technology; quality of life; motion based; intervention
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motion based intervention (Experimental): To examine whether the activity of virtual cycling contributes to the improvement of quality of life for individuals with cognitive impairment
  Interventions: Other: Motion based - Virtual cycling
- No intervention (No Intervention): no intervention for this group

INTERVENTIONS:
Other: Motion based - Virtual cycling — To examine whether the activity of virtual cycling contributes to the improvement of quality of life for individuals with cognitive impairment. (Intervention study)
  Arms: Motion based intervention

SUMMARY:
The aging population is growing in Sweden and worldwide, highlighting the urgent need to address their needs using available societal resources. In Swedish nursing homes, about 80,000 people reside, 70% of whom have cognitive impairments, and many are physically inactive. Cognitive impairment negatively impacts daily activities and quality of life, and is the most common reason for moving from home to a nursing home. Methods to meet these individuals' needs must be developed to motivate physical, cognitive, and social activation, aiming to improve the quality of life for older people with cognitive impairments.

Movement-based interactive technology is a type of welfare technology that uses a virtual environment to stimulate activity. Virtual cycling is one example, where the individual pedals a stationary bike while watching a self-chosen interactive film. Virtual cycling thus includes multiple elements such as physical activation and cognitive and social stimulation. Previous research has shown virtual cycling to be a promising method for older adults with cognitive impairments. Few nursing homes have used this method, but a pilot project (unpublished) at nursing home for people with dementia, the investigators observed positive effects on the residents' quality of life. Virtual cycling has only been evaluated in three small international research studies, none of which have examined the impact on participants' quality of life. Therefore, the project's aim is to evaluate whether virtual cycling can improve quality of life and the physical, social, and cognitive activity abilities of older people with cognitive impairments.

1. Does virtual cycling contribute to an improved quality of life for older people with cognitive impairment?
2. How do residential staff and research assistants perceive the impact of virtual cycling on the physical, social, and cognitive abilities, as well as the quality of life, of older people with cognitive impairment?
3. What experiences do residential staff and research assistants have regarding the opportunities and obstacles for implementing virtual cycling?

DETAILED DESCRIPTION:
The project includes two studies;

Study 1) The Intervention Study

A Randomized Controlled Trial (RCT) study with a quantitative design. Approximately 60-80 people will be included in the intervention study and randomized into either the intervention group or the control group. The cycling intervention involves cycling twice a week for 8 weeks, with each session lasting about 40 minutes.The intervention will be carried out at the nursing home where the participant resides.

Measurement instruments will be used where participants will answer questions and perform physical tests. Observation instruments and questionnaires with questions concerning the participants will be answered by residential staff and research assistants. Information regarding necessary medications and Body mass index will be obtained from the participants' health and medical records from the municipality.

Analysis Pre- and post-measurements will be conducted.The results from the measurements will be statistically analyzed and the outcomes compared between the intervention group and the control group. The results will be analyzed according to the intention-to-treat principle, meaning that all participants' results will be analyzed regardless of whether they completed the intervention or not. The results will also be analyzed per protocol, meaning that only individuals who completed the intervention (16 cycling sessions) will be included in the analysis.

Description of the Virtual Cycling Intervention The intervention to be carried out involves the participant cycling on a stationary bike while an interactive film plays on a large-screen Television. The films allow the participant to cycle through various landscapes, cities, etc., and the participant can choose the film based on their previous experiences and interests, to create a motivating activity. Participants will perform the activity individually, together with a research assistant. The research assistant is a specialist nurse assistant (specially trained in the field of dementia or welfare technology) who is well-versed in working with people with dementia and works daily with this client group. The research assistant will be active during the activity and stimulate the participant to talk about what they see and experience while cycling to enhance the participant's cognitive and social activity abilities.

Study 2) The Interview Study

After the intervention (study 1) is completed, a qualitative study will be conducted using semi-structured interviews with residential staff and research assistants. The interview guide includes questions about participants' daily activities before, during, and after the intervention, changes in quality of life, participants' experiences of the intervention, and thoughts on using the virtual bike in the residence. Approximately 25-30 residential staff/research assistants are planned to be interviewed until saturation is reached. All interviews will be conducted by a doctoral student and will take about 45 minutes each. The interviews will be recorded and transcribed verbatim.The interviews with the residential staff will take place approximately 2-4 weeks after the end of the cycling intervention. The research assistants will be interviewed approximately 2-4 weeks after all cycling interventions have been completed.

Analysis The interviews and questionnaire responses will be analyzed inductively, where meaning units, condensed meaning units, codes, and categories form themes that describe the entire material. The themes will be illustrated with quotes. The analyses will be conducted using the software NVivo 12. Some of the interviewed participants will be selected to discuss the analyzed results with the doctoral student and a researcher at one occasion. This procedure increases the validity of the interview study.

ELIGIBILITY:
Study 1)

Inclusion Criteria:

* age more than 65
* resides in a nursing home
* cognitive impairment measured by MMSE, scoring <24 points on the MMSE.

Exclusion Criteria:

* Individuals who cannot provide their own informed consent will be excluded, in consultation with their relatives/guardians.
* Individuals who cannot do the movement to the cycle

Study 2)

Inclusion Criteria:

* no age limits
* the residential staff should have worked closely with the participant in the intervention study for three months before the intervention began.
* the residential staff should have worked closely with the participant during the duration of the intervention study (16 sessions).
* the residential staff should have participated once when the participant conducted the cycling intervention, as the staff member being interviewed.

Exclusion Criteria:

- residential staff who are not assessed to understand and speak Swedish to an extent that allows the interview to be conducted will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life- Quality of Life in Late-Stage Dementia | 10 weeks
  Quality of Life in Late-Stage Dementia (QUALID) is a proxy instrument and assesses observable quality of life in dementia. The QUALID includes eleven questions about observed behavior and mood (smiling, appearing sad, crying, irritable, etc.) that assess quality of life in dementia on a five-point Likert scale. The result of the test is scored between 11-55 points, where lower scores indicate a higher quality of life. It will be conducted two times, approximately 1-2 weeks before and after the intervention, for both the treatment group and the control group. The required time for the test is 15 minutes.

SECONDARY OUTCOMES:
Quality of life- EuroQol-5 Dimensions-5 Levels | 10 weeks
  EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) measures quality of life and will be used as both a self-assessment instrument and a proxy instrument. The instrument consists of two parts, with the first part containing five health dimensions: mobility, daily activities, self-care, pain/discomfort, and anxiety/depression. The EQ-5D-5L is an extension of the original EQ-5D with expanded response options, including five statements indicating whether an individual has "no," "slight," "moderate," "severe," or "extremely severe" problems within the dimensions. In the second part of the instrument, the individual's general health is assessed using a visual analog scale (VAS).
  It will be conducted two times, approximately 1-2 weeks before and after the intervention, for both the treatment group and the control group. The required time for the test is 15 minutes.
Behavioral and psychological symptoms- The Neuropsychiatric Inventory | 10 weeks
  The Neuropsychiatric Inventory (NPI) measures behavioral and psychological symptoms through observation in individuals with dementia. Through observations, the presence and severity of 12 symptoms are assessed, such as agitation, depression, anxiety, apathy, and motor restlessness. The instrument rates the presence (Likert scale, 1-4 points) and severity (Likert scale, 0-3 points) of the various symptoms. The frequency and severity scores are multiplied to produce a total score ranging from 0 to 144 points, with higher scores indicating more severe symptoms.
  It is a proxy instrument and it will be conducted two times, approximately 1-2 weeks before and after the intervention, for both the treatment group and the control group. The required time for the test is 15 minutes.
Physical test- The Timed Chair Stand Test | 10 weeks
  The Timed Chair Stand Test (TCST), measures strength in the lower extremities. The participant is to perform ten chair rises from a chair (height 45 cm). The participant must stand up fully and sit down completely each time. The outcome measure is the time in seconds, with a longer time indicating a higher risk of falls in older adults.
  It will be conducted two times, approximately 1-2 weeks before and after the intervention, for both the treatment group and the control group. The required time for the test is 15 minutes.
Physical test- The Timed Up and Go | 10 weeks
  The Timed Up and Go (TUG), assesses and measures mobility and proactive balance. The participant is to rise from a seated position in an armchair, walk 3 meters, turn around, walk back, and sit down. The time taken to complete this task is measured. The outcome measure is the time in seconds, with a longer time indicating a higher risk of falls in older adults.
  It will be conducted two times, approximately 1-2 weeks before and after the intervention, for both the treatment group and the control group. The required time for the test is 15 minutes.
Cognitive test- The Mini-Mental State Examination | 10 weeks
  The Mini-Mental State Examination (MMSE), is a screening instrument for cognitive impairment. The instrument consists of 20 questions (maximum 30 points) and assesses cognitive functions, such as orientation, memory, language, and visuospatial ability. Lower points indicate more cognitive difficulties. Indication of dementia is has cut-off of <24 points (out of 30 points).
  It will be conducted two times, approximately 1-2 weeks before and after the intervention, for both the treatment group and the control group. The required time for the test is 30 minutes.

OTHER OUTCOMES:
Use of medication | 12 weeks
  Medication that the participant takes to counteract behavioral and psychological symptoms associated with dementia. Information about the quantity of necessary medication taken over a period of one month is collected from the participants health journal before the intervention begins and once after the intervention ends, covering a month's consumption period.
Health data- Body Mass Index | 10 weeks
  Body Mass Index (BMI) is a measure that calculates whether a person is underweight, normal weight, or overweight. BMI is taken from the participants health journal once before the intervention begins and once after the intervention ends.
Number of falls | 24 weeks
  Information gather from medical records regarding the number of times the participants of this study has fallen within the two months before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Matérne, Principal Investigator — Örebro University, Sweden
Locations (1):
- School of behavioural, social and legal sciences, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
We could share on other researchers request.

REFERENCES:
- [Background] de Souto Barreto P, Morley JE, Chodzko-Zajko W, H Pitkala K, Weening-Djiksterhuis E, Rodriguez-Manas L, Barbagallo M, Rosendahl E, Sinclair A, Landi F, Izquierdo M, Vellas B, Rolland Y; International Association of Gerontology and Geriatrics - Global Aging Research Network (IAGG-GARN) and the IAGG European Region Clinical Section. Recommendations on Physical Activity and Exercise for Older Adults Living in Long-Term Care Facilities: A Taskforce Report. J Am Med Dir Assoc. 2016 May 1;17(5):381-92. doi: 10.1016/j.jamda.2016.01.021. Epub 2016 Mar 21. PMID 27012368
- [Background] Moyle W, Jones C, Murfield J, Draper B, Beattie E, Shum D, Thalib L, O'Dwyer S, Mervin CM. Levels of physical activity and sleep patterns among older people with dementia living in long-term care facilities: A 24-h snapshot. Maturitas. 2017 Aug;102:62-68. doi: 10.1016/j.maturitas.2017.05.015. Epub 2017 May 30. PMID 28610686
- [Background] Dove E, Astell AJ. The Use of Motion-Based Technology for People Living With Dementia or Mild Cognitive Impairment: A Literature Review. J Med Internet Res. 2017 Jan 11;19(1):e3. doi: 10.2196/jmir.6518. PMID 28077346
- [Background] D'Cunha NM, Isbel ST, Frost J, Fearon A, McKune AJ, Naumovski N, Kellett J. Effects of a virtual group cycling experience on people living with dementia: A mixed method pilot study. Dementia (London). 2021 Jul;20(5):1518-1535. doi: 10.1177/1471301220951328. Epub 2020 Aug 21. PMID 32820955
- [Background] Marinus N, Hansen D, Feys P, Meesen R, Timmermans A, Spildooren J. Cycling: how can we activate care-dependent older adults with a mild cognitive impairment? Disabil Rehabil Assist Technol. 2023 Aug;18(6):896-903. doi: 10.1080/17483107.2021.1936665. Epub 2021 Jun 8. PMID 34102092
- [Background] Zorz S, Dellaire S, Reilly K, Wilson-Sanchez J, Rodriguez RA, Campbell TM. Reminiscence-tied cycling technology in long-term care: A feasibility study. J Am Geriatr Soc. 2021 Oct;69(10):2987-2990. doi: 10.1111/jgs.17307. Epub 2021 Jun 5. No abstract available. PMID 34089262
- [Background] Weiner MF, Martin-Cook K, Svetlik DA, Saine K, Foster B, Fontaine CS. The quality of life in late-stage dementia (QUALID) scale. J Am Med Dir Assoc. 2000 May-Jun;1(3):114-6. PMID 12818023
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204